CLINICAL TRIAL: NCT06506201
Title: Legs Dysmetria in Total Hip Replacement: Does Hip Approacches and Navigation Decrease the Risk?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0005971
Record Dates: First submitted 2024-06-17; First posted 2024-07-17 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- direct anterior approach with navigation assistance (Experimental): Patients treated surgically with total hip arthroplasty (direct anterior approach) with navigation assistance.
  Interventions: Device: Velys hip navigation
- direct anterior approach without navigation assistance (Active Comparator): Patients treated surgically with total hip arthroplasty (direct anterior approach) without navigation assistance.
  Interventions: Procedure: Standard of care
- lateral direct approach with navigation assistance (Experimental): Patients treated surgically with total hip arthroplasty (lateral direct approach) with navigation assistance.
  Interventions: Device: Velys hip navigation
- lateral direct approach without navigation assistance (Active Comparator): Patients treated surgically with total hip arthroplasty (lateral direct approach) without navigation assistance.
  Interventions: Procedure: Standard of care
- postero-lateral approach with navigation assistance (Experimental): Patients treated surgically with total hip arthroplasty (postero-lateral approach) with navigation assistance.
  Interventions: Device: Velys hip navigation
- postero-lateral approach without navigation assistance (Active Comparator): Patients treated surgically with total hip arthroplasty (postero-lateral approach) without navigation assistance.
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Device: Velys hip navigation — Computer assisted surgery
  Arms: direct anterior approach with navigation assistance; lateral direct approach with navigation assistance; postero-lateral approach with navigation assistance
Procedure: Standard of care — surgery without navigation
  Arms: direct anterior approach without navigation assistance; lateral direct approach without navigation assistance; postero-lateral approach without navigation assistance

SUMMARY:
The purpose of this study is to collect clinical and radiological data from the case series of patients surgically treated with total hip arthroplasty at the Rizzoli Orthopaedic Institute.

The primary objective is to evaluate in terms of safety and efficacy the reduction of legs dysmetria and proper acetabular cup inclination intraoperatively when comparing anterior, direct lateral, and postero-lateral hip approaches conducted via traditional or navigation-assisted surgery.

The secondary objectives of the study are to evaluate, by comparing navigation-assisted and non-navigation-assisted hip approaches, intraoperatively the correct positioning of the prosthesis by analyzing the acetabular cup version; surgical timing; and number of intraoperative radiographs taken. In addition, the accuracy of preoperative planning will be assessed and a clinical evaluation performed during a follow-up of one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 and 80 years;
2. Signs and symptoms of hip osteoarthritis (pain intensity of at least 6 points of visual analogic scale pain - 0-10 scale in the previous week);
3. Radiographic signs of hip osteoarthritis (Grade 3-4 according to Tonnis classification);

Exclusion Criteria:

1. Patients unable to express consent;
2. Patients undergoing previous ipsilateral hip surgery;
3. Patients undergoing lower limb surgery to be treated in the previous 12 months;
4. Patients with malignant neoplasms;
5. Patients with rheumatic diseases;
6. Patients with uncontrolled diabetes;
7. Patients with uncontrolled thyroid metabolic disorders;
8. Patients abusing alcoholic beverages, drugs or medications;
9. Body Mass Index > 35;
10. Pregnant and/or fertile women.
11. Pain intensity less than 6 points in accordance with the visual analogic scale scale.
12. Patients with the presence of excessive deformity resulting from acetabular or femoral head dysplasia
13. Patients who have already undergone total hip arthroplasty surgery on the affected hip.
14. Previous extensive surgery of the reference joint (osteotomy around the hip, open or arthroscopic osteochondroplasty for femoral-acetabular conflict).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Legs dysmetria in millimeters calculated in anteroposterior x-rays | Intraoperatory
  Legs lenght dysmetria in total hip replacement surgery

SECONDARY OUTCOMES:
Cup orientation in grade° calculated in anteroposterior x-rays | Intraoperatory
  Cup orientation in total hip replacement surgery

CONTACTS AND LOCATIONS:
Overall Officials: Federico Raggi, MD, Principal Investigator — Isitituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No